CLINICAL TRIAL: NCT03993665
Title: Use of Multiparametric Magnetic Resonance Imaging in the Management of Head and Neck Cancer: a Prospective Analysis
Brief Title: Use of Multiparametric MRI in the Management of Head and Neck Cancer: a Prospective Analysis
Status: Active, not recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, head of department, AZ Sint-Jan AV
Other Study IDs: B049201838067
Record Dates: First submitted 2019-02-13; First posted 2019-06-21 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer; Multiparametric MRI; Cervical Lymph Node; Bone Invasion; Tumour Relapse; Treatment Response
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- affected: All patients with a histologically confirmed squamous cell carcinoma in the head and neck region
- control: Whartin tumour or pleomorphic adenoma of the parotid gland without malignant transformation

SUMMARY:
The investigators aim to validate specific MRI parameters that could improve diagnostic accuracy of metastatic cervical lymph nodes in patients with a squamous cell carcinoma in the head and neck region. Moreover, we aim to explore specific MRI parameters that could improve diagnostic accuracy of bone invasion and tumour relapse, as well as predict treatment response and survival in this target population.

DETAILED DESCRIPTION:
Background: The locoregional control rates in patients with advanced head and neck cancer remain suboptimal. Accurate diagnosis of metastatic cervical lymph nodes, bone invasion, or tumour relapse in a previously irradiated or operated field remains challenging. Technological advances in magnetic resonance imaging (MRI) enable to quantify diffusion and perfusion of the tumour and its surrounding tissues, which could improve diagnostic performance. Moreover, they could provide additional information about radiation and/or chemotherapeutic efficiency in an individual patient.

Objectives: The investigators aim to validate specific MRI parameters that could improve diagnostic accuracy of metastatic cervical lymph nodes in patients with a squamous cell carcinoma in the head and neck region. Moreover, we aim to explore specific MRI parameters that could improve diagnostic accuracy of bone invasion and tumour relapse, as well as predict treatment response and survival in this target population.

Methods: In this trial, a validation cohort will be recruited in a prospective manner, to validate the MRI parameters that showed clinically acceptable discriminant value based on the retrospective study. The values of the selected MRI parameters will be calculated in metastatic lymph nodes of the affected group, for comparison with their values measured in the lymph nodes of a prospectively recruited control group, comprising patients who require the same standardized MRI protocol for evaluation of a Whartin tumour or pleomorphic adenoma of the parotid gland without malignant transformation, and in whom both the parotid gland lesion and the cervical lymph node are surgically removed for histological confirmation. All included patients of the 'affected group' will also undergo a preoperative positron emission tomography-computed tomography (PET-CT), according to international guidelines, and will preferably receive a multiparametric MRI at 3, 6, 12, 24, 36, 48 and 60 months post treatment as part of routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a pretreatment multiparametric MRI according to a standardized protocol
* Histopathologically proven SCC in the HN region (affected group)
* Histopathologically proven Whartin tumour or pleomorphic adenoma in the HN region without malignant transformation (control group)
* Patients in whom a or multiple clearly distinguishable cervical lymph node(s) can be observed radiologically, and which can be correlated unambiguously with the pathology report

Exclusion Criteria:

* not fulfilling abovementioned criteria
* thyroid or skin cancer
* considerable artefact on MRI
* previously surgery, irradiation or chemotherapy in the HN region

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Histopathologically proven SCC in the HN region (affected group)
  - Histopathologically proven Whartin tumour or pleomorphic adenoma in the HN region without malignant transformation (control group)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
discriminatory value of MRI perfusion curve between tumoural and non-tumoural cervical lymph nodes | preoperative
  MRI parameters will be considered validated if they enable differentiation between a metastatic cervical lymph node and a non-tumoural lymph node, as based on the final pathology report as the 'gold standard'
discriminatory value of MRI ADC value between tumoural and non-tumoural cervical lymph nodes | preoperative
  MRI parameters will be considered validated if they enable differentiation between a metastatic cervical lymph node and a non-tumoural lymph node, as based on the final pathology report as the 'gold standard'
discriminatory value of MRI D value between tumoural and non-tumoural cervical lymph nodes | preoperative
  MRI parameters will be considered validated if they enable differentiation between a metastatic cervical lymph node and a non-tumoural lymph node, as based on the final pathology report as the 'gold standard'

SECONDARY OUTCOMES:
discriminatory value of perfusion curve between bone invasion and no bone invasion | preoperative
  MRI parameters will be considered validated if they enable differentiation between tumoural bone invasion and no bone invasion, as based on the final pathology report as the 'gold standard'
discriminatory value of predefined perfusion curve between post-therapeutic sequelae and tumour relapse | follow-up until 5 years postoperative
  MRI parameters will be considered validated if they enable differentiation between post-therapeutic sequelae and tumour relapse, as based on the final pathology report as the 'gold standard'
predictive value of the MRI parameter Ktrans for treatment outcome | end of adjuvant radiochemotherapy (approx 10 weeks postoperative)
  predictive value of MRI parameters for treatment outcome, measured through tumoural response at therapy end based on the RECIST criteria
predictive value of predefined Ktrans for overall and disease-free survival | postoperative follow-up at 3, 6, 12, 24, 36,48 and 60 months
  predictive value of MRI parameters for treatment outcome, measured through tumoural response at therapy end based on the RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (1):
- Division of Maxillofacial Surgery, Department of Surgery, AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No